CLINICAL TRIAL: NCT01275625
Title: A Multicenter, Open Label Study Of Maraviroc, Zidovudine And Lamivudine Twice Daily For The Treatment Of Antiretroviral Naïve HIV-Infected Patients With R5 HIV-1 In Russia
Brief Title: Combivir And Maraviroc In Antiretroviral Naive Subjects In Russia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4001101
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-01

CONDITIONS: HIV
Keywords: maraviroc; naive; hiv; zidovudine; lamivudine; combivir; Clade A
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Single arm study of combivir and maraviroc for 48 weeks
  Interventions: Drug: HIV therapy

INTERVENTIONS:
Drug: HIV therapy — Combivir one tablet BD with maraviroc 300mg BD for 48 weeks
  Other Names: Selzentry, Celsentri

SUMMARY:
One hundred subjects in Russia will be treated with a combination of Combivir (zidovudine and lamivudine) and maraviroc as their first line HIV therapy. The aim is to assess the efficacy and safety of this combination in a Russian population of patients.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* R5 HIV infection on screening tropism test.
* Viral load >1,000 copies/mL.
* Never previously treated with anti-HIV medicines.

Exclusion Criteria:

* Previously treated with anti-HIV medicines.
* Hepatitis B co-infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Russia (8):
  - Regional Center on AIDS and Infectious Diseases Prophylaxis and Control, Krasnoyarsk
  - Federal scientific and methodological center on AIDS prophylaxis and control, Moscow
  - Moscow regional center on AIDS and infectious diseases prophylaxis and control, Moscow
  - Regional Center on AIDS and Infectious Diseases Prophylaxis and Control, Nizhny Novgorod
  - Saint-Petersburg Center on AIDS and Infectious Diseases Prophylaxis and Control, Saint Petersburg
  - Federal State Institution Republican clinical infectious hospital of Roszdrav, Saint Petersburg
  - Smolensk Center on AIDS and infectious diseases prophylaxis and control, Smolensk
  - Volgograd Regional Center on AIDS and Infectious Diseases Prophylaxis and Control, Volgograd

REFERENCES:
- [Derived] Lewis ME, Jubb B, Simpson P, Lopatukhin A, Kireev D, Bobkova M, Craig C, van der Ryst E, Westby M, Butler SL. Highly prevalent Russian HIV-1 V3-loop sequence variants are susceptible to maraviroc. Antivir Chem Chemother. 2021 Jan-Dec;29:20402066211025156. doi: 10.1177/20402066211025156. PMID 34160290
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001101&StudyName=Combivir%20And%20Maraviroc%20In%20Antiretroviral%20Naive%20Subjects%20In%20Russia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This report presents results of a 48 week study conducted at 8 centers in Russia. A total of 98 subjects were enrolled in the study; however, one site was closed and data from this site was deemed unusable, thus in total 77 subjects were included in the analysis.
Pre-assignment Details: Treatment naïve Human Immuno Deficiency Virus (HIV) infected participants aged 18 years at screening were enrolled. Participants were required to meet all eligibility criteria prior to randomization into the study.
Groups:
- Maraviroc+Combivir: All participants received Maraviroc (300 milligram [mg] twice daily) in combination with Combivir (fixed dose combination of zidovudine 300 mg and lamivudine 150 mg)
Period: Overall Study
Arm/Group | Maraviroc+Combivir
Started | 77
Treated | 77
Completed | 64
Not Completed | 13
Not completed — Death | 1
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 4
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Maraviroc+Combivir
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immuno Deficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) Load <50 Copies/Milliliter (mL) at 48 Weeks.
Description: Participants' responder status at Week 48 was assessed according to Missing, discontinuation= Failure (MDF) algorithm. This algorithm treats all participants with HIV 1 RNA data missing at the time of interest or discontinuation of study drug as failures or non responders.
Time Frame: 48 weeks
Population: Full Analysis Set (FAS) Population included those participants who had taken at least 1 dose of the study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maraviroc+Combivir
Number analyzed (Participants) | 77
Percentage of participants | 77.92 [68.01 to 87.84]

2. Secondary Outcome: Virologic Response: Percentage of Participants With Plasma HIV-1 RNA Load <50 Copies/mL at Post-baseline Visits.
Description: Participants' responder status at Week 48 was assessed according to MDF algorithm. This algorithm treats all participants with HIV 1 RNA data missing at the time of interest or discontinuation of study drug as failures or non responders.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 20, Week 24, Week 36 and Week 48
Population: FAS Population included those participants who had taken at least 1 dose of the study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc+Combivir
Number analyzed (Participants) | 77
Percentage of participants
  Baseline (N= 77) | 0.00
  Week 4 (N= 77) | 7.79
  Week 8 (N= 75) | 26.67
  Week 12 (N= 76) | 48.68
  Week 20 (N= 73) | 78.08
  Week 24 (N= 73) | 83.56
  Week 36 (N= 68) | 89.71
  Week 48 (N= 65) | 92.31

3. Secondary Outcome: Virologic Response: Percentage of Participants With Plasma HIV-1 RNA Load < 400 Copies/mL at Post-baseline Visits.
Description: as for outcome 2
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 20, Week 24, Week 36 and Week 48
Population: FAS Population included those participants who had taken at least 1 dose of the study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Maraviroc+Combivir
Number analyzed (Participants) | 77
Percentage of participants
  Baseline (N= 77) | 0.00
  Week 4 (N= 77) | 41.56
  Week 8 (N= 75) | 72.00
  Week 12 (N= 76) | 89.47
  Week 20 (N= 73) | 91.78
  Week 24 (N= 73) | 91.78
  Week 36 (N= 68) | 97.06
  Week 48 (N= 65) | 95.38

4. Secondary Outcome: Virologic Response: Rate of Virologic Failure at Week 48.
Description: Virologic failure defined as: failure to achieve a reduction from baseline in HIV 1 RNA ≥ 0.5 log10 copies /mL by the second viral load determination (unless viral load was below the lower limit level of quantification [LLOQ]); or a ≥ 0.5 log10 increase from nadir in HIV 1 RNA after achieving a HIV 1 RNA reduction from BL >0.5 log10 copies/mL; or a HIV 1 RNA level of >1000 copies/mL after having achieved a HIV 1 RNA level below LLOQ. Participants with Time to loss of virologic response (defined by level of <50 copies/mL) failure were classified as rebounders or non-responders.
Time Frame: 48 weeks
Population: FAS Population included those participants who had taken at least 1 dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Maraviroc+Combivir
Number analyzed (Participants) | 77
Participants
  Responders | 60
  Rebounders | 1
  Non-response | 15
  Death | 1
  Discontinued before Week 48 due to Adverse Events | 4
  Discontinued before Week 48 for other reasons | 9

5. Secondary Outcome: Immunological Response at Week 48: Absolute Change From Baseline in Absolute Cluster of Differentiation 4 (CD4)
Description: Immunological Response was summarized using absolute change from Baseline to Week 48 in absolute CD4+ cell count
Time Frame: Week 48
Population: FAS Population included those participants who had taken at least 1 dose of the study drug.
Measure: Mean (Standard Deviation); unit: cells/microliter (cells/mcL)
Arm/Group | Maraviroc+Combivir
Number analyzed (Participants) | 64
cells/microliter (cells/mcL) | 165.53 (163.65)

6. Secondary Outcome: Immunological Response at Week 48: Percentage Change From Baseline in Absolute Cluster of Differentiation 4 (CD4)
Description: Immunological Response was summarized using percentage change from Baseline to Week 48 in absolute CD4+ cell count
Time Frame: Week 48
Population: FAS Population included those participants who had taken at least 1 dose of the study drug.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Maraviroc+Combivir
Number analyzed (Participants) | 64
Percent | 8.07 (7.14)

7. Secondary Outcome: Immunological Response at Week 48: Absolute Change From Baseline in Absolute Cluster of Differentiation 8 (CD8)
Description: Immunological Response was summarized using absolute change from Baseline to Week 48 in absolute CD8+ cell count.
Time Frame: Week 48
Population: FAS Population included those participants who had taken at least 1 dose of the study drug.
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | Maraviroc+Combivir
Number analyzed (Participants) | 64
cells/mcL | -112.96 (361.85)

8. Secondary Outcome: Immunological Response at Week 48: Percentage Change From Baseline in Absolute Cluster of Differentiation 8 (CD8)
Description: Immunological Response was summarized using percentage change from Baseline to Week 48 in absolute CD8+ cell count.
Time Frame: Week 48
Population: FAS Population included those participants who had taken at least 1 dose of the study drug.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Maraviroc+Combivir
Number analyzed (Participants) | 64
Percent | -8.59 (9.28)

9. Secondary Outcome: Immunological Response at Week 48: Change From Baseline in Absolute Cluster of Differentiation 4 (CD4)/ Cluster of Differentiation 8 (CD8) Ratio.
Description: Immunological Response was summarized using absolute change from Baseline to Week 48 in absolute CD4+/ CD8+ ratio.
Time Frame: Week 48
Population: FAS Population included those participants who had taken at least 1 dose of the study drug.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Maraviroc+Combivir
Number analyzed (Participants) | 64
Ratio | 0.33 (0.90)

10. Secondary Outcome: Number of Participants With Genotypic Resistance.
Description: The viral genotypes were captured at Baseline and at treatment failure or Early termination and any resistance-associated mutations summarized descriptively at Week 48 for the Nucleotide reverse transcriptase inhibitors (NRTIs), and non-NRTIs (NNRTIs)drug classes.
Time Frame: Screening to Week 48 or Time of treatment Failure
Population: All participants who discontinued therapy early or who reached Week 48 with sufficient plasma HIV 1 RNA for analysis (500 copies/mL) were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Maraviroc+Combivir
Number analyzed (Participants) | 77
Participants
  Participants with genotype reported | 8
  Participants with Emergent NRTI mutations | 5

11. Secondary Outcome: Number of Participants With HIV-1 RNA Tropism Status Using Genotyping Assay at Screening and at the Time of Virologic Failure.
Description: Change in tropism were summarized at the time of treatment failure or Early Termination (note: this was performed for participants with viral load > 400 copies/mL only).
Time Frame: Screening to Week 48 or Time of treatment Failure
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Maraviroc+Combivir
Number analyzed (Participants) | 77
Participants
  Tropism change (n= 8) | 0
  Reduced Maraviroc susceptibility (n= 3) | 0

ADVERSE EVENTS:
Time Frame: Baseline to follow-up period (28 days after the last dose of study)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Maraviroc+Combivir
Serious Adverse Events (participants affected / at risk) | 2/77
Other Adverse Events (participants affected / at risk) | 51/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc+Combivir (N=77)
Anemia (Blood and lymphatic system disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc+Combivir (N=77)
Anemia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Abnormal faeces (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 2
Fatigue (General disorders) | 1
Malaise (General disorders) | 8
Performance status decreased (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 3
Chronic sinusitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 9
Respiratory tract infection viral (Infections and infestations) | 5
Salpingo-oophoritis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Vaginitis bacterial (Infections and infestations) | 1
Viral rhinitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 6
Blood pressure increased (Investigations) | 2
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Hypoaesthesia (Nervous system disorders) | 1
Intercostal neuralgia (Nervous system disorders) | 1
Neuritis cranial (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Drug dependence (Psychiatric disorders) | 1
Neurogenic bladder (Renal and urinary disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Nail psoriasis (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Cows milk free diet (Surgical and medical procedures) | 1
Angina pectoris (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Amylase increased (Investigations) | 1
Heart rate increased (Investigations) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Cervicobrachial syndrome (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Essential hypertension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.